CLINICAL TRIAL: NCT01303705
Title: Phase Ib Study of Monoclonal Antibody to OX40, Cyclophosphamide (CTX) and Radiation in Patients With Progressive Metastatic Prostate Cancer After Systemic Therapy
Brief Title: Anti-OX40, Cyclophosphamide (CTX) and Radiation in Patients With Progressive Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH&S IRB 10-088
Record Dates: First submitted 2010-11-09; First posted 2011-02-25 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Prostate Cancer; Cancer of the Prostate; Prostate Cancer
Keywords: progressive metastatic prostate cancer; cancer of the prostate; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cyclophosphamide - Cohort 1 (Experimental): Cyclophosphamide 300 mg/m2 IV on Day 1; Radiation Therapy 8.0 Gy in 1 fraction to a maximum of three bone metastatic deposits will be administered on Day 4 of treatment; Anti-OX40 will be administered intravenously at 0.4 mg/kg on days 4, 6 and 8.
  Interventions: Drug: Anti-OX40; Radiation: Radiation; Drug: Cyclophosphamide
- Cyclophosphamide - Cohort 2 (Experimental): Cyclophosphamide 600 mg/m2 IV on Day 1; Radiation Therapy 8.0 Gy in 1 fraction to a maximum of three bone metastatic deposits will be administered on Day 4 of treatment; Anti-OX40 will be administered intravenously at 0.4 mg/kg on days 4, 6 and 8.
  Interventions: Drug: Anti-OX40; Radiation: Radiation; Drug: Cyclophosphamide
- Cyclophosphamide - Cohort 3 (Experimental): Cyclophosphamide 900 mg/m2 IV on Day 1; Radiation Therapy 8.0 Gy in 1 fraction to a maximum of three bone metastatic deposits will be administered on Day 4 of treatment; Anti-OX40 will be administered intravenously at 0.4 mg/kg on days 4, 6 and 8.
  Interventions: Drug: Anti-OX40; Radiation: Radiation; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Anti-OX40 — Anti-OX40 will be administered intravenously at 0.4 mg/kg on days 4, 6 and 8 of the study. The total anti-OX40 dose will be reconstituted in 100 ml 0.9% saline and infused over no more than 60 minutes intravenously. A single-use non-pyrogenic durapore membrane low protein binding filter (e.g.: Braun 1.2 micron air eliminating filter or equivalent) shall be used to filter the study product in the line between infusion bag and patient.
  Other Names: MEDI6469
Radiation: Radiation — 8.0 Gy in 1 fraction to a maximum of three bone metastatic deposits will be administered on Day 4 of treatment. Imaging such as bone scan, MRI, CT scan, or radiograph must identify the target lesion as consistent with metastatic disease. Any bone lesion that is inducing pain or where there may be a clinical concern for potential pathological fracture will be selected over asymptomatic lesions.
  Other Names: Rx
Drug: Cyclophosphamide — CTX will be administered on day 1 (Friday only) at a dose determined by cohort assignment. The drug should be diluted per institutional standards. An added dose of IV fluids may help prevent bladder toxicity. In this protocol, CTX will be administered intravenously over 30 - 60 minutes.
  Other Names: CTX; Cytoxan

SUMMARY:
This clinical trial will examine a novel combination of anti-OX40 to induce proliferation of memory and effector T cells in conjunction with cyclophosphamide (CTX) and radiation to induce tumor antigen release with the overall goal of promoting an immune response against prostate cancer.

DETAILED DESCRIPTION:
A Phase Ib trial design will be employed in patients with metastatic PC who have failed prior androgen ablation and docetaxel. CTX will be administered also on Day 1. All patients will receive RT (800 cGy in a single fraction) to up to 3 bone metastatic sites on Day 4 in the AM. Anti-OX40 at 0.4 mg/kg IV will be given on days 4, 6 and 8. The timing of CTX, RT and anti-OX40 are based on the pre-clinical models and the observation that the synergies of CTX and RT are reduced when they are given more than one week after anti-OX40 and are maximized when given within 3 days of starting anti-OX40. The proposed radiation dose is commonly used to palliate bone pain in PC and generally will not induce significant cytopenias. The CTX dose will be escalated in successive cohorts of 3 - 6 patients to assure patient safety. The dose levels of CTX will be 300, 600 and 900 mg/m2 intravenously in the initial stage of the study. The range of CTX doses is commonly used in general oncology practice and is not expected to induce prolonged myelosuppression, although transient cytopenias are likely. Concurrent CTX and RT has been well-tolerated at much higher dose-intensities than the investigators are proposing (52-54), thus the investigators are not expecting significant adverse events from the combination before anti-OX40. As a safety consideration, the investigators are not giving CTX and RT on the same day as a high proportion of men with prostate cancer have bone metastases in the pelvis. RT to the pelvis could cause radiation cystitis that would be exacerbated by the metabolites of CTX (e.g., acrolein) that can accumulate in the bladder in the 24-36 hours after administration. After the dose-escalation portion of the trial then up to 20 additional patients can enroll in the study at the maximum tolerated CTX dose if clinical responses are seen, for a maximum total of 37 patients using a Simon two-stage design (see Section 10 for details).

The main clinical objective of the trial will be to characterize toxicity and estimate the response rate of the combination of anti-OX40, CTX and RT. Both radiographic and PSA responses will be followed. RECIST will be used for radiographic assessment and a significant PSA response will be defined as a 50% or greater decrease from baseline measured at 3 and 6 weeks after the start of treatment based on the PCWG2 guidelines (55).

Patients will enroll consecutively to each cohort assuming no dose-limiting toxicities. Three patients will be treated per cohort and if there are no dose-limiting toxicities, then enrollment to the next cohort can begin. If a dose-limiting toxicity is encountered in the first three patients in any cohort, then an additional three patients will be enrolled in that cohort.* This dosing strategy will allow for a three-fold escalation of CTX.

The main hypothesis of this study is that CTX and RT will induce tumor breakdown providing a source of antigen for self-vaccination and anti-OX40 will amplify CD8-mediated effector responses across a broad spectrum of prostate cancer antigens resulting in further regression of prostate cancer. The investigators predict that anti-OX40 will not increase circulating or intratumoral Treg, and this should help to further augment immune responses.

*For the dose escalation portion of the study, the first 2 patients in any cohort can be treated on consecutive weeks. If there are no Dose Limiting Toxicities, then the third patient can begin treatment 28 days after the second patient has completed anti-OX40. If the third patient has no DLT, then the next cohort can open 28 days after the third patient has completed anti-OX40. If a DLT occurs with patient 3 in any cohort, then up to 3 more patients will enroll to the same cohort at a frequency of one patient every 28 days after the previous patient has completed anti-OX40 assuming no DLT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with measurable or evaluable metastatic adenocarcinoma of the prostate. Either histologic or cytologic diagnosis is acceptable
2. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 (Appendix A.)
3. Age 18 years old or above
4. Laboratory values (performed within 28 days prior to enrollment) as follows:

   * WBC ≥ 2000/microlitre
   * Serum creatinine < 1.5 X upper limit of laboratory normal
   * Hgb > 8g/dl (patients may be transfused to reach this level)
   * Platelets > 100,000 cells/mm3
   * Total bilirubin < 1.5 X upper limit of laboratory normal, unless due to Gilbert's disease
   * AST (SGOT) and ALT (SGPT) < 2.5 X upper limit of laboratory normal
   * Alkaline phosphatase < 2.5 X upper limit of laboratory normal (If alkaline phosphatase > 2.5 X upper limit of laboratory normal due to bone metastases, then patient is eligible.)
   * HIV 1 and 2 antibody Negative
   * Hepatitis B surface antigen Negative
   * Hepatitis C antibody Negative
   * PSA > 2 ng/ml
   * Testosterone < 50 ng/ml
5. Confirmed radiographic and/or PSA progression (using PCWG2 definitions) after at least one androgen ablation regimen and docetaxel.Patients who refuse docetaxel chemotherapy or who are not candidates for docetaxel are eligible to enroll.
6. At least one bone metastatic lesion amenable to radiation
7. Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand the investigational nature of the study and the risks associated with the therapy
8. No active bleeding
9. No clinical coagulopathy (INR < 1.5, PT < 16 seconds, PTT < 38 seconds)
10. Anticipated lifespan greater than 12 weeks
11. Patients on LHRH agonists or bisphosphonates prior to study enrollment should continue these medications without change

Exclusion Criteria:

1. Active infection.
2. Active autoimmune disease.
3. Previous treatment with mouse monoclonal antibodies
4. Need for chronic maintenance oral steroids.
5. Active brain metastatic disease. Patients with treated brain metastases with surgery, gamma-knife radiosurgery or radiation and stable for at least 4 weeks and off steroids are eligible.
6. Any medical or psychiatric condition that in the opinion of the PI would preclude compliance with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10-14 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | The MTD will be assessed according to the dose escalation schema (timeframe is not specific for MTD assessment - it is based on enrollment)*
  The primary objective of this trial is to determine the maximum tolerated dose (within the range expected to induce anti-tumor and immunological effects) of CTX administered in combination with radiation and anti-OX40 in men with metastatic castrate- and chemotherapy-resistant prostate cancer.

SECONDARY OUTCOMES:
Immune and Clinical Responses | Days 11, 18, 25 and 39
  Secondary objectives are as follows:
  1. Determine the effect of anti-OX40, CTX and radiation on circulating numbers and phenotypes of CD4 and CD8 T cells.
  2. Measure the proliferation and activity of effector and memory T cells after CTX, radiation and anti-OX40.
  3. Perform exploratory studies of cellular and humoral immune responses against prostate cancer cell lines.
  4. Estimate the response rate of the regimen that includes the highest dose of CTX determined to be safe.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan D Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No